CLINICAL TRIAL: NCT05815225
Title: Neuroinflammation Markers in Subjects With Psychotic Symptoms
Acronym: NEUROINPS17
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROINPS17
Record Dates: First submitted 2023-02-01; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Neuroinflammatory Response; Psychosis
Keywords: psychosis; cytokines; chemokines; endocannabinoid system
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood collection at the 3 cut-off points. 18 mL of blood will be obtained in EDTA tubes (K2, K3). A tube will be used to obtain plasma, which will be frozen within an hour and a half after extraction. It is necessary to perform the centrifuge at 4º, obtaining as many aliquots of 500 microliters (at least 3) as possible. The remainder less than 500 ul will be stored in a single aliquot. The second tube will be used to obtain white blood cells according to the protocol established by the Biobank together with the research group. Cryopreservation will be done at -70ªC in the IBIMA Biobank.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: subjects from mental health unit: Subjects with active psychotic symptoms at the time of recruitment, attended at the Mental Health Clinical Management Unit of the Regional University Hospital of Malaga (Spain) and admitted to the Mental Health Hospitalization Unit. In turn, within this group, a cross-classification will be established according to the evolutionary staging of the disease, the concomitant presence of major affective symptoms and the consumption of substances in the weeks prior to admission.
- B: subjects with induced psychoses: Subjects with psychotic symptoms, diagnosed with a substance-induced psychotic episode, already recruitedand previously characterized.
- C: control group: Control group of volunteers extracted from the general population, without psychotic symptoms orsubstance use disorders.

SUMMARY:
The main objective of the study is to measure the plasma and intracellular levels of several neuroinflammation markers (including cytokines and chemokines) and the endocannabinoid system in subjects presenting psychotic symptoms, initially recruited in a Mental Health Hospitalization Unit, and in different stages of their disease.

To this end, we will evaluate and clinically characterize a cohort of patients who present active psychotic symptoms at the time of recruitment, and comparing it with a control group with similar sociodemographic characteristics. We will also compare our sample with a smaller sample previously recruited from patients with substance use and psychotic symptoms. Within our cohort of patients with psychotic symptomatology we will distinguish in turn affective psychoses from non-affective psychoses, on the one hand; and induced and non-induced psychosis by drug consumption, on the other. We will also classify patients based on whether they are experiencing the first episode of their illness or a relapse.

This is an observational, longitudinal and prospective study. 3 blood draws will be performed from the subjects included in the study: the first, in the first 48 hours of hospital admission; the second, in the 48 hours prior to discharge; and the third, 6 months after discharge. The rater team will be composed of senior psychiatrists and training psychiatrists. The sample will be composed of subjects with psychotic symptoms who come from the Mental Health Clinical Management Unit of the Regional University Hospital of Malaga. Each patient enrolled in this study will undergo a clinical evaluation (psychiatric diagnostic interview and psychometric scales). From the plasma and white blood cells of the blood sample, the biochemical levels of the inflammatory mediators will be determined. Demographic, clinical, and biochemical data will be assessed and analysed using statistical programmes.

DETAILED DESCRIPTION:
The main objective of the study is to measure the plasma and intracellular levels of several neuroinflammation markers (including cytokines and chemokines) and the endocannabinoid system in subjects presenting psychotic symptoms, initially recruited in a Mental Health Hospitalization Unit, and in different clinical and evolutive stages of their disease.

To this end, we will evaluate and clinically characterize a cohort of patients who present active psychotic symptoms at the time of recruitment, and comparing it with a control group with similar sociodemographic characteristics. We will also compare our sample with a smaller sample previously recruited from patients with substance use and induced psychotic symptoms. Within our cohort of patients with psychotic symptomatology we will distinguish in turn affective psychoses from non-affective psychoses, on the one hand; and induced and non-induced psychosis by drug consumption, on the other. We will also classify patients based on whether they are experiencing the first episode of their illness or a relapse.

This study has two parts. The first one is an observational, longitudinal and prospective study. 3 blood draws will be performed from the subjects included in the study (group A of participants, see below): the first, in the first 48 hours of hospital admission; the second, in the 48 hours prior to discharge; and the third, 6 months after discharge. The sample will be composed of subjects with psychotic symptoms who come from the Mental Health Clinical Management Unit of the Regional University Hospital of Malaga. Each patient enrolled in this study will undergo a clinical evaluation (psychiatric diagnostic interview and psychometric scales). Figure 1 represents this study.

The second one is a cross-sectional study in which we will compare measurements made in group A participants with a previously recruited sample of patients with substance-induced psychosis (group B, see below) and a sample of healthy, non-psychotic controls (group C, see below).

The rater team will be composed of senior psychiatrists and training psychiatrists. From the plasma and white blood cells of the blood sample, the biochemical levels of the inflammatory mediators will be determined. Demographic, clinical, and biochemical data will be assessed and analyzed using statistical programs.

This study will be carried out in a brief psychiatric hospitalization unit located in the city of Malaga (Andalusia, Spain) and has 42 beds for a catchment area of approximately 500.000 inhabitants. This unit is part of the Mental Health care system within the Andalusian Health Service, which provides universal health coverage to all people living in the autonomous community. The mental health department of the hospital also comprises other units such as two community mental health centers, one day center, one medium- and long-stay ward (30 beds), one child and adolescent mental health unit, an intensive community treatment team, a care team for first episodes of psychosis, and an eating disorders unit.

The process of collecting clinical data and extracting peripheral blood will be carried out as follows:

1. Signature of the informed consent and appointment for evaluation process.
2. Venous blood collection at the 3 cut-off points listed above. 18 mL of blood will be obtained in EDTA tubes (K2, K3). A tube will be used to obtain plasma, which will be frozen within an hour and a half after extraction. It is necessary to perform the centrifuge at 4º, obtaining as many aliquots of 500 microliters (at least 3) as possible. The remainder less than 500 ul will be stored in a single aliquot. The second tube will be used to obtain white blood cells according to the protocol established by the Biobank together with the research group. Cryopreservation will be done at -70ªC in the IBIMA Biobank.
3. Apply clinical evaluation instruments (see section assessment instruments).
4. The plasma evaluation of the concentrations of the molecular species differences: N-acylethanolamines, 2-acylglycerols and cytokines (including chemokines) will be carried out in the laboratory of the Civil Hospital of Málaga.
5. The samples will be processed and stored in the Biobank of the Civil Hospital of Málaga.

Both qualitative and quantitative descriptive statistics will be used to characterize the sample that has participated in the study as demographic and diagnostic information.

Demographics. Comparisons between groups or hypothesis testing will be made by the Chi Square test (χ2) or Fisher's exact formula in the case of qualitative variables and by Student's T statistic or analysis of variance (ANOVA) in the case of quantitative variables. Non parametric test (Mann-Whitney test and Kruskal-Wallis) will be used if the distributions not follow normality. For all hypothesis testing a probability p<0.05 will be considered significant.

Clinical and biochemical data. The results will be expressed with the number of subjects and respective percentage, as well as by means of the means and standard deviations (SD). Statistical significations will be determined by Fisher's exact test or chi-square test and Student's t-test (Welch correction with unequal variances). For comparison, between the one- and two-way groups, analyses of variance followed by the post hoc test of multiple comparisons (Bonferroni test) will be used. Correlation analyses will be performed through Pearson's coefficient. In addition, the receiver operating characteristics (ROC) will be analyzed taking into account the area under the curve (AUC) and these will be used to generate regression models which in turn will create predictors.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men and women) with diagnostic criteria for psychotic episode, affective episode with psychotic symptoms, or substance-induced psychotic episode, according to DSM and ICD criteria.
* Age from 18 to 65 years.
* Informed consent.

Exclusion Criteria:

* Severe cognitive alterations that do not allow the application of diagnostic instruments.
* Infectious diseases [Laboratory prophylaxis (HIV, Hepatitis B, C)].
* Not speaking the Spanish language fluently.
* History of head trauma with loss of consciousness, stroke, or CNS disease.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A sample of subjects with psychotic symptoms (divided into several clinical subgroups) at different stages of their disease will be compared with another sample of patients with psychotic symptoms already recruited previously and a control group of people from the community without psychiatric pathology or substance use.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Level of biomakers 1 | Week 1
  Levels of endocannabinoids and neuroinflammation mediators (cytokines and chemokines) in subjects with active psychotic symptoms
Level of biomakers 2 | Week 1-8
  Levels of endocannabinoids and neuroinflammation mediators (cytokines and chemokines) in subjects with active psychotic symptoms
Level of biomakers 3 | Week 22-26
  Levels of endocannabinoids and neuroinflammation mediators (cytokines and chemokines) in subjects with active psychotic symptoms
Changes from Baseline level of biomarkers at 6 months | Week 1 and Week 22-26
  Changes from Baseline level of biomarkers at 6 months

SECONDARY OUTCOMES:
Rate of phenotype characteristics and clinical symptoms | Week 22-26
  Rate of phenotype characteristics and clinical symptoms of patients with psychotic symptoms, including affective and non-affective psychoses and induced and not induced by drug consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Mayoral-Cleríes, MD, Study Chair — Hospital Regional de Malaga
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Spain